CLINICAL TRIAL: NCT00058994
Title: An Evaluation of Safety and Efficacy of Anecortave Acetate Versus Placebo in Patients With Subfoveal Choroidal Neovascularization Due to Exudative Age-related Macular Degeneration
Brief Title: An Evaluation of Safety and Efficacy of Anecortave Acetate Versus Placebo in Patients With Subfoveal CNV Due to Exudative AMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-02-29
Record Dates: First submitted 2003-04-15; First posted 2003-04-16 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2008-08

CONDITIONS: Macular Degeneration; Maculopathy, Age-Related
Keywords: AMD; anecortave acetate; wet AMD; age-related macular degeneration; Macular Degeneration; Maculopathy, Age-Related; Age-Related Maculopathies; Age-Related Maculopathy; Maculopathies, Age-Related
MeSH Terms: conditions — Macular Degeneration | interventions — anecortave acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: anecortave acetate

SUMMARY:
The purpose of this study is to demonstrate that anecortave acetate is superior to placebo in maintenance of visual acuity at the 12- and 24-month visits.

ELIGIBILITY:
Patients at least 50 years of age, of any race, and either sex with a clinical diagnosis of exudative AMD and a primary or recurrent subfoveal CNV lesion in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-03; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Investigators, Principal Investigator — Alcon Research
Locations (1):
- South America, Fort Worth, Texas, United States